CLINICAL TRIAL: NCT01891747
Title: A Phase I/II Study of High-dose L-methylfolate in With Combination Temozolomide and Bevacizumab in Recurrent High Grade Glioma.
Brief Title: A Phase I Study of High-dose L-methylfolate in Combination With Temozolomide and Bevacizumab in Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Stephen Clark, MD, Assistant Professor of Neurology, Neuro-oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC NEU 1308
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Malignant Glioma
Keywords: gliomas
MeSH Terms: conditions — Glioma | interventions — Bevacizumab; Temozolomide; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-methylfolate with Bevacizumab & Temozolomide (Experimental): 28-day cycle, dose levels L-methylfolate: Phase I 15 mg (once a day) 30 mg (15 mg twice a day) 60 mg (30 mg twice a day) 90 mg (45 mg twice a day) Phase II will use the MTD of L-methylfolate daily with bevacizumab & temozolomide.
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Bevacizumab — bevacizumab at 10mg/kg IV every 14 days (Phase I & phase II)
Drug: Temozolomide — 150 mg/m2/day for a 5-day regimen per month (Phase I & Phase II)
Dietary Supplement: Vitamin C — 250 mg vitamin C once a day (oral) - Phase I & Phase II

SUMMARY:
This is a Phase I/II non-randomized prospective study of high-dose L-methylfolate in combination with bevacizumab and temozolomide in patients with recurrent high-grade glioma. The primary objective of this phase II trial is to determine whether the addition of high-dose L-methylfolate to bevacizumab and temozolomide therapy improves progression-free survival (PFS) compared to previously reported results.

DETAILED DESCRIPTION:
The phase I part of the study will be completed to determine the Maximum Tolerated Dose (MTD) of high-dose L-methylfolate in combination with bevacizumab at 10mg/kg IV every 14 days, a 5-day regimen per month of temozolomide at 150 mg/m2/day and a 250 mg tablet of vitamin C. Dose escalation will involve 3 patients treated at each dose level of L-methylfolate (15mg, 30 mg, 60 mg or 90 mg), and the MTD will be confirmed by expansion of 3 additional patients. It is anticipated that 6 to 15 patients will be enrolled in the phase 1 part of the study. Patients will continue treatment until disease progression. Once the MTD of L-methylfolate has been determined, patients enrolled at a lower dose level may increase L-methylfolate dose to the MTD dose, per investigator discretion.

The phase II part of the study will consist of patients taking the MTD of L-methylfolate daily in combination with bevacizumab at 10 mg/kg IV every 14 days, a 5-day regimen per month of temozolomide at 150 mg/m2/day and a 250 mg tablet of vitamin C. There will be 32 patients treated in the Phase II study and the patients will continue treatment until progression. The 6 patients treated at the MTD cohort in Phase

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignant glioma (anaplastic oligodendroglioma, anaplastic astrocytoma, anaplastic oligoastroctyoma or glioblastoma). Patients must have genetically confirmed Isocitrate dehydrogenase I (IDH1) wild-type tumor.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as greater than or equal to 5 mm. Patients can have non-measurable disease if they have had recent surgery for radiographic progression.
* Patients can have been treated with standard therapy for high grade glioma, including surgical resection, chemoradiation with temozolomide, adjuvant temozolomide and bevacizumab. Patients can have received experimental therapy for high grade glioma.
* Patients must be 18 years of age or older.
* Patients may not be breast-feeding a child.
* Patients must have a Karnofsky Performance Score of greater than or equal to 60 percent.
* Patients must have normal organ and marrow function as defined below:

leukocytes greater than or equal to 3,000/milliliter (mcL) absolute neutrophil count greater than or equal to 1,500/mcL platelets greater than or equal to 100,000/mcL total bilirubin within normal institutional limits Aspartate transaminase (serum glutamic oxaloacetic transaminase)Alanine transaminase (Serum Glutamic Pyruvate Transaminase) less than or equal to 2.5 times institutional upper limit of normal Creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60/mL/min 1.73 m2 for patients with creatinine levels above institutional normal

* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast. Patients with prior malignancies must be disease-free for greater than or equal to 3 years.
* The effects of high-dose L-methylfolate on the developing human fetus at the recommended therapeutic dose are unknown, but, there is evidence that folic acid can be protective against neural tube defects. However, there is some concern that folate supplementation can increase the incidence of autism, and thus women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately. All women will have pregnancy testing performed prior to entering the trial.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patients must be able to tolerate MRIs. CT scans can NOT be substituted for MRI in this study.
* Patients on therapeutic warfarin or enoxaparin are eligible.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (greater than grade I) due to agents administered more than 4 weeks earlier.
* Patients with genetically confirmed IDH1-mutated tumor.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to folic acid.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, stage II hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because high-dose folic acid has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with high-dose folic acid breastfeeding should be discontinued if the mother is treated with high-dose folic acid.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with high-dose folic acid. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (Phase I) | every 4 weeks, 28-day cycle, up to 6 months
Progression-free survival (Phase II) | On treatment to disease progression or death for any reason, up to 12 months
  Disease progression is defined as either radiological or clinical/neurological progression (whichever occurs first), PFS is the time interval between the date of starting treatment and the date of disease progression or death, whichever comes first. If neither event has been observed, then the patient is censored at the date last documented to be free of progression. Progression-free and overall survival will be summarized non-parametrically using the method of Kaplan and Meier with standard errors based on Greenwood's formula.

SECONDARY OUTCOMES:
Objective Response (Phase I) | every 8 weeks, up to 6 months
  Response will be determined by neurologic examination and contrast-enhanced MRI initially after 8 weeks and then subsequently prior to every other cycle based on the Response Assessment in Neuro-Oncology criteria (RANO).
Number of patients with each worst-grade toxicity. (Phase I) | every 4 weeks (28-day cycle), up to 6 months
  To determine the safety profile of high-dose L-methylfolate (15mg, 30 mg, 60 mg or 90 mg) in combination with bevacizumab and temozolomide in patients with recurrent high-grade glioma as determined by number of patients with each worst grade toxicity using the Common Terminology Criteria for Adverse Events 4.0, 1 = mild through 5 = death.
Overall Survival (Phase II) | on study to date of death, up to 12 month
  median overall survival and time to survival in patients treated with L-methylfolate in combination with temozolomide and bevacizumab. The Duration of survival is the time interval between the date of starting treatment and the date of death. Patients still alive will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Clark, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/